CLINICAL TRIAL: NCT06922123
Title: Behavioural and Neurophysiological Reactions During Tactile Stimulation in Patients Suffering From Disorders of Consciousness (DoC)
Brief Title: Tactile Stimulation in Disorders of Consciousness (DoC)
Acronym: TACTILE-DOC
Status: Not yet recruiting | Type: Observational
Sponsor: Anna Estraneo (Other)
Collaborators: University of Liege (Other)
Responsible Party: Sponsor-Investigator, Anna Estraneo, MD Neurologist Senior researcher, Fondazione Don Carlo Gnocchi Onlus
Organization: Fondazione Don Carlo Gnocchi Onlus (Other)
Other Study IDs: TACTILE-DOC
Record Dates: First submitted 2025-03-26; First posted 2025-04-10 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Disorders of Consciousness
Keywords: Tactile stimulation; Disorders of Consciousness; Behavioural evaluation; Neurophysiological evaluation; Pleasant touch stimulation
MeSH Terms: conditions — Consciousness Disorders | interventions — Neurophysiological Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with Disorders of Consciousness (DoC): All patients with disorders of consciousness who are consecutively admitted to the participating centers of the study will be enrolled with a diagnosis of disorders of consciousness based on the CRS-R scale, with an age ≥18 years and a time since the event ≥ 28 days.
  Interventions: Behavioral: Tactile stimulation; Device: Neurophysiological Monitoring with SedLine

INTERVENTIONS:
Behavioral: Tactile stimulation — Patients will undergo a resting-state EEG and fNIRS recording, followed by the administration of the SECONDs scale. Tactile stimulation will then be performed on eight areas of the body (internal and external forearms, palms and backs of the hands on both sides) using six different stimuli categorized as pleasant, neutral, or unpleasant. Stimuli will be applied manually in randomized blocks. EEG and fNIRS data will be recorded before, during, and after stimulation. Behavioural responses will be evaluated through video analysis by independent raters. The session will last approximately 90 minutes.
Device: Neurophysiological Monitoring with SedLine — SedLine is a non-invasive neurophysiological monitoring device used to record the brain's electrical activity (EEG) through frontal electrodes. In this study, SedLine is employed to measure resting-state and stimulus-evoked cortical responses in patients with disorders of consciousness (DoC), in combination with functional near-infrared spectroscopy (fNIRS). The EEG signals are used to assess changes in neural activity before, during, and after tactile stimulation with various affective valences (pleasant, neutral, unpleasant). This combined multimodal approach enhances the understanding of sensory processing and cortical reactivity in patients with impaired consciousness.
  Other Names: SedLine EEG Monitor; Masimo SedLine

SUMMARY:
The aim of this project is to evaluate the behavioural and neurophysiological responses to pleasant touch in patients with disorders of consciousness (DoC) and to determine whether these responses are related to the level of consciousness. Specifically, the study aims to:

1. explore the relationship between pleasant tactile stimulation and behavioural and neurophysiological responses in patients with DoC;
2. determine whether behavioural responses to pleasant touch stimulation correlate with the level of consciousness;
3. assess whether behavioural responses vary depending on the valence of the stimulus (pleasant, neutral, or unpleasant);
4. examine neurophysiological responses to tactile stimulation using functional near-infrared spectroscopy (fNIRS), and evaluate whether brain activation patterns are associated with behavioural responses;
5. improve diagnostic accuracy in patients with DoC by exploring the value of somatosensory responses in distinguishing unresponsive wakefulness syndrome (UWS) from minimally conscious state (MCS) or conscious patients;
6. explore the potential usefulness of implementing this type of stimulation within rehabilitation programs to support better recovery of consciousness.

DETAILED DESCRIPTION:
Patients will be enrolled at the participating centers and included in the study only after at least two evaluations using the Coma Recovery Scale-Revised (CRS-R), in order to ensure a stable diagnosis of the level of consciousness.

At the beginning of the protocol, non-invasive fNIRS optodes will be placed on the patient's forehead using a frontal headband, and 15 minutes of resting-state brain activity will be recorded. The Simplified Evaluation of CONsciousness Disorders (SECONDs) will then be administered to assess the patient's level of consciousness, followed by the tactile stimulation protocol.

The tactile stimulation protocol involves 8 areas of the body (anterior and posterior forearm, palm and back of the hand, on both right and left sides) and 6 stimuli grouped into three categories: pleasant objects (makeup brush, plush fabric), neutral objects (sponge, rubber fabric), and unpleasant objects (dishnet, hairbrush). Each stimulus is mounted on a 10 cm wooden stick attached to a cork base. Each stimulation lasts 15 seconds and is manually administered using light circular movements over an area of approximately 5 cm² at a speed of 5 cm/s, following a randomized sequence. A 10-second rest period will be provided between stimulations. Patients will receive three distinct blocks of stimulation: unpleasant stimuli (first block), pleasant stimuli (second block), and neutral stimuli (third block), with the block order randomized across participants. After each block, the SECONDs will be re-administered to detect any changes in the level of consciousness. An additional 15-minute resting-state fNIRS recording will follow the stimulation phase.

All sessions will be video-recorded to allow two independent experimenters to evaluate behavioural responses (e.g., facial expressions, vocalizations, body movements, and emotional reactions such as crying, smiling, or grimacing) and compare the effects of different stimulations. At the end of the session, fNIRS optodes will be removed.

The entire experimental procedure will last approximately 90 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a disorder of consciousness (DoC), as determined by repeated Coma Recovery Scale-Revised (CRS-R) assessments;
* Age ≥ 18 years;
* Time since acute event ≥ 28 days.
* Written informed consent obtained from the legal representative

Exclusion Criteria:

* Presence of large craniectomy that may interfere with fNIRS signal acquisition;
* Unstable clinical conditions (e.g., respiratory insufficiency, fever, status epilepticus);
* Fractures, paralysis, lesions, or muscular atrophy that prevent proper tactile stimulation of the specified body areas;
* Absence of informed consent from the legal representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with DoC who are consecutively admitted to the participating centers of the study
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
SECONDs Scale Total Score Pre- and Post-Tactile Stimulation | Day 1 (immediately before and after each stimulation block)
  Consciousness level will be assessed using the Simplified Evaluation of CONsciousness Disorders (SECONDs) scale at baseline and after each stimulation block (pleasant, neutral, unpleasant). Score changes will be recorded to evaluate short-term effects of stimulation valence.
Behavioral Response Scores During Tactile Stimulation (Video Coding) | Day 1 (during stimulation phase)
  Video recordings will be rated by two independent observers for presence and intensity of facial expressions, vocalizations, body movements, and emotional indicator. A composite behavioral response score will be computed for each stimulus type.
Hemodynamic Response Changes to Tactile Stimuli Measured by fNIRS | Day 1 (before, during, and after stimulation)
  Changes in oxyhemoglobin (HbO) and deoxyhemoglobin (HbR) concentrations will be measured using functional near-infrared spectroscopy (fNIRS) over frontal areas. Signal changes will be analyzed by stimulus valence and correlated with behavioural responses.
Cortical Activation Patterns During Tactile Stimulation (EEG - SedLine) | Day 1 (before, during, and after stimulation)
  EEG signals will be recorded via SedLine during the full session. Changes in spectral power (e.g., delta, theta, alpha, beta bands) will be analyzed across stimulation blocks to determine cortical reactivity to pleasant, neutral, and unpleasant touch.

SECONDARY OUTCOMES:
Change in Simplified Evaluation of CONsciousness Disorders (SECONDs) Score From Baseline to Post-Stimulation | Day 1 (pre and post each of the 3 stimulation blocks)
  The Simplified Evaluation of CONsciousness Disorders (SECONDs) is a clinical scale used to quantify the patient's consciousness level. It consists of six behavioural items with a total score ranging from 0 to 8, where higher scores represent better levels of consciousness. The Simplified Evaluation of CONsciousness Disorders (SECONDs) scores will be submitted before and after each stimulation block and will be compared to determine short-term modulation of consciousness level to explore the value of somatosensory processing responses of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Estraneo, MD, Principal Investigator — Fondazione Don Gnocchi; Olivia Gosseries, PhD, Professor, Principal Investigator — University of Liege

IPD SHARING:
Plan to Share IPD: Yes
IPD collected throughout the trial (SECONDs, video recordings outcomes, fNIRS, EEG data).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From the first patient recording data until the last patient.